CLINICAL TRIAL: NCT03226015
Title: Autologous Oral Mucosa With Amniotic Membrane Transplantation for Limbal Stem Cell Deficiency: Clinical and Immunohistochemical Study
Brief Title: Autologous Oral Mucosa Transplantation for Limbal Stem Cell Deficiency
Status: Completed | Type: Observational
Sponsor: Klinikum Chemnitz gGmbH (Other)
Collaborators: Institute of Anatomy TU Dresden (Unknown)
Responsible Party: Principal Investigator, Katrin Engelmann, Head of Ophthalmology, Klinikum Chemnitz gGmbH
Other Study IDs: EK-BR-64/15-1
Record Dates: First submitted 2017-07-13; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Limbal Stem-cell Deficiency
Keywords: Limbal Stem-cell Deficiency; Oral mucosa transplantation; Amniotic membrane; Mesenchymal stem cells
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — oral mucosa tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PURPOSE: To report clinical and histochemical results of oral mucosa graft transplantation in eyes with limbal stem cell deficiency.

DESIGN: Prospective observational study.

METHODS: 32 eyes of 27 patients with limbal stem cell deficiency underwent direct oral mucosa graft transplantation with amniotic membrane transplantation with a mean follow-up of 19 months. Clinical course of the disease including emergency surgeries, planned curative procedures, conjunctival inflammation, acute inpatient treatment and best corrected visual acuity were assessed at 3 months postoperatively and at last follow up visit. The unneeded parts of oral mucosa graft were analyzed immunohistochemically with staining for mesenchymal stem cell markers and pericytes (CD 90, CD 146, CD 166, CD 31, CD 68, protein gene product).

ELIGIBILITY:
Inclusion Criteria:

* limbal stem cell deficiency at least in one eye
* undergoing oral mucosa with amniotic membrane transplantation
* obtained written informed consent

Exclusion Criteria:

* no written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with oral mucosa with amniotic membrane transplantation in Klinikum Chemnitz 2015-2017
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
change in number of acute surgeries | baseline, 3 months after oral mucosa transplantation; through study completion, an average of 19 months
change in days of acute inpatient treatment | baseline, 3 months after oral mucosa transplantation; through study completion, an average of 19 months

SECONDARY OUTCOMES:
change in number of curative surgical procedures after oral mucosa transplantation | baseline, 3 months after oral mucosa transplantation; through study completion, an average of 19 months
change in conjunctival inflammation | baseline, 3 months after oral mucosa transplantation; through study completion, an average of 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Engelmann, PhD, Principal Investigator — Klinikum Chemnitz